CLINICAL TRIAL: NCT04631978
Title: Analysis of Retinochoroidal Vasculature in Underweight Women Using Optical Coherence Tomography Angiography
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Aslı Çetinkaya Yaprak, Principal Investigator, Akdeniz University
Other Study IDs: 19102017-15/4-184
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Cachexia; Underweight
MeSH Terms: conditions — Cachexia; Thinness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Underweight: Comprehensive ophthalmologic examination
  Interventions: Diagnostic Test: Comprehensive ophthalmologic examination
- Control: Comprehensive ophthalmologic examination
  Interventions: Diagnostic Test: Comprehensive ophthalmologic examination

INTERVENTIONS:
Diagnostic Test: Comprehensive ophthalmologic examination — Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and optical coherence tomography angiography imaging.

SUMMARY:
Cachectic patients and controls undergoing a comprehensive ophthalmologic examination. The imaging of all subjects is undertaken using a commercial OCTA device with a scan rate of 70,000 A-scans/s, scan beam wavelength of 840 ± 10 nm and bandwidth of 45 nm. All measurements are performed between 10:00 and 12:00 on the same day. The OCTA images are independently graded and assessed by two retinal specialists. The software automatically segmented these full-thickness retinal scans into the superficial and deep inner retinal vascular plexuses, outer retina, and choriocapillaris (CC). The vascular density in the superficial and deep retinal vascular zones is calculated automatically by the software, and the foveal avascular zone (FAZ) and foveal density (FD) are also automatically determined. Choroidal thickness is calculated manually by two retinal specialists, and the average value was used.

DETAILED DESCRIPTION:
Cachectic patients and controls undergoing a comprehensive ophthalmologic examination, including the measurements of best-corrected visual acuity (BCVA), refractive error (KR-8900; Topcon, Tokyo, Japan), intraocular pressure (IOP, Full Auto Tonometer TX-F; Topcon), axial length (AL, Lenstar LS 900, Haag-Streit AG, Switzerland), slit lamp examination of the anterior segment, dilated fundus examination, and OCTA imaging (Optovue RTVue XR 100 Avanti, Freemont, California, USA) are included in the study. To calculate BMI, height is measured using a standard anthropometric tape (Bioplus Stature Meter, model number IND/09/2005/815), and a certified electronic weighing scale (model number Omron HN-283) is used to measure weight.

According to the national guidelines, the patients are classified into two underweight groups: Group 1 consisting of those with a BMI of <17.00 kg/m2 and Group 2 comprising those with a BMI of 17.00 to 18.49 kg/m2. The control group is formed with individuals with a normal BMI (18.50 to 24.99 kg/m2).

The right eye of each participant is included in the study. If the right eye meets any of the exclusion criteria, then the left eye is selected for the sample. The inclusion criteria for the patient group is being underweight (BMI < 18.50 kg/m2). The exclusion criteria for all groups are as follows: refractive error >+3.0 diopters (D) or <-3.0 D spherical equivalent; poor image quality <60 due to unstable fixation; IOP > 21 mm Hg; longer AL (>25 mm); pre-existing ophthalmic pathologies; prior ocular surgery; and a systemic chronic disease that can cause underweight or retinopathy, such as cancer, malnutrition, and diabetes mellitus.

OCTA

The imaging of all subjects is undertaken using a commercial OCTA device with a scan rate of 70,000 A-scans/s, scan beam wavelength of 840 ± 10 nm and bandwidth of 45 nm. This device can perform 70 000 A-scans/s per second to acquire volumes of 304 × 304 A-scans. All measurements are performed between 10:00 and 12:00 on the same day.

To evaluate the vascular structures, 6×6 mm OCTA software is used. The split-spectrum amplitude decorrelation angiography (SSADA) algorithm is performed in all participants. The images of poor quality (signal strength index (SSI) < 8) with either significant motion artifact or incorrect segmentation are excluded. The OCTA images are independently graded and assessed by two retinal specialists. The software automatically segmented these full-thickness retinal scans into the superficial and deep inner retinal vascular plexuses, outer retina, and choriocapillaris (CC). The vascular density in the superficial and deep retinal vascular zones is calculated automatically by the software, and the foveal avascular zone (FAZ) and foveal density (FD) are also automatically determined. The same software also calculates the flow index rates in a central circular zone of 3.144 mm² in the outer retina and CC segments. Choroidal thickness is calculated manually by two retinal specialists, and the average value was used.

ELIGIBILITY:
Inclusion Criteria:

* Underweight (BMI < 18.50 kg/m2).

Exclusion Criteria:

* refractive error >+3.0 diopters (D) or <-3.0 D spherical equivalent;
* poor image quality <60 due to unstable fixation
* IOP > 21 mm Hg
* longer AL (>25 mm)
* pre-existing ophthalmic pathologies
* prior ocular surgery
* a systemic chronic disease that can cause underweight or retinopathy, such as cancer, malnutrition, and diabetes mellitus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population includes a convenience sampling from the patients admitted to outpatient clinic between June 2020 and August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Choriocapillaris flow area | 10 minutes
  Choriocapillaris flow area assessed with optical coherence tomography angiography

SECONDARY OUTCOMES:
Subfoveal choroidal thickness | 10 minutes
  Subfoveal choroidal thickness assessed with optical coherence tomography angiography
Vessel density | 10 minutes
  Vessel density assessed with optical coherence tomography angiography
Foveal avascular zone | 10 minutes
  Foveal avascular zone assessed with optical coherence tomography angiography
Subfoveal central macular thickness | 10 minutes
  Subfoveal central macular thickness assessed with optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Çentinkaya Yaprak, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No